CLINICAL TRIAL: NCT00622544
Title: A Prospective Study of Microalbuminuria in Untreated Boys With Alport Syndrome
Acronym: MA
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 0707M11722
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2017-09

CONDITIONS: Alport Syndrome; Kidney Disease
Keywords: Microalbuminuria; Proteinuria
MeSH Terms: conditions — Nephritis, Hereditary; Kidney Diseases; Proteinuria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Each urine sample will be assayed for albumin, total protein and creatinine. The following definitions will be used:
  * Microalbuminuria: urine albumin:creatinine ratio (ACR) > 30 mcg/mg, on 3 consecutive measurements spaced one month apart
  * Overt proteinuria: urine protein:creatinine ratio (UPC) > 0.2 mg/mg, on 3 consecutive measurements spaced one month apart
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of the Microalbuminuria in Untreated Boys with Alport Syndrome study is to gather information about critical clinical time points such as when patients with small amounts of protein (microalbuminuria) in their urine progress to larger amounts (overt proteinuria). Large amounts of protein in the urine is often an early sign of kidney disease.

Information needs to be collected in boys who are not taking medications known as angiotensin converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) in order to obtain accurate data about the length of time between the onset of microalbuminuria and the start of overt proteinuria. This new information will give physicians a better understanding of how to treat patients with Alport syndrome.

The information we gather by conducting this study will aid in planning future clinical trials because the identification of time points in disease progression, such as microalbuminuria and overt proteinuria, could reduce the time necessary to show a clinical benefit of a new treatment option.

The study has been approved by the University of Minnesota's Institutional Review Board.

DETAILED DESCRIPTION:
Study Aims

1. To determine the average ages of onset of microalbuminuria and overt proteinuria in untreated boys with Alport syndrome
2. To determine the average duration of microalbuminuria before transition to overt proteinuria in untreated boys with Alport syndrome

This study does not involve treatment and is anticipated to last 3-5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alport syndrome, confirmed by skin biopsy, kidney biopsy, or molecular genetic analysis
* Diagnosis of Alport syndrome, based on presence of hematuria and confirmed diagnosis of Alport syndrome in a first-degree relative
* Male gender
* Absence of overt proteinuria, defined as urine protein:creatinine ratio less than 0.2 mg/mg
* Subject is not currently receiving treatment with an angiotensin converting enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB)

Exclusion Criteria:

* Female gender
* Presence of overt proteinuria
* Current treatment with ACEI or ARB
* End-stage kidney disease (on dialysis or kidney transplant recipient)

Max Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population is comprised of approximately 30 males ranging in age from 0 - 18 at the time of enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2007-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifford E Kashtan, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Observational Study: no Arms - One Group: Observational study of urine albumin and protein excretion in untreated boys with X-linked Alport syndrome
Period: Overall Study
Arm/Group | Observational Study: no Arms - One Group
Started | 44
Completed | 35 (35)
Not Completed | 9

BASELINE CHARACTERISTICS:
Groups:
- Observational Study: no Arms - One Group: Observational study of urine albumin and protein excretion in untreated boys with Alport syndrome
Arm/Group | Observational Study: no Arms - One Group
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.9 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Developing Microalbuminuria During Study Period
Description: number of subjects developing microalbuminuria during study period
Time Frame: 2007-2009
Measure: Count of Participants; unit: Participants
Groups:
- Observational Study: no Arms - One Group: Boys less than 18 years of age with a confirmed diagnosis of Alport syndrome
Arm/Group | Observational Study: no Arms - One Group
Number analyzed (Participants) | 35
Participants | 35

2. Secondary Outcome: Number of Subjects Developing Proteinuria During the Study Period
Description: number of subjects developing proteinuria during the study period
Time Frame: 2007-2009
Measure: Count of Participants; unit: Participants
Arm/Group | Observational Study: no Arms - One Group
Number analyzed (Participants) | 35
Participants | 35

ADVERSE EVENTS:
Time Frame: 2007-2009
Arm/Group | Observational Study: no Arms - One Group
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No